

NCT03986216

October 26, 2020

For each of the surveyed questions (scaled from 1-5 with 1 representing the no satisfied and 5 as very satisfied), we will calculate the mean and standard deviation, with a focus on identifying scores < 3/5.

We will use single and paired T-tests to determine the effects of PT experience and the number of training sessions on participant satisfaction, respectively.

We will use the repeated measure of ANOVA to test whether the training session number plays a role in the hand function as primarily measured by Box and Blocks Test and the other secondary measures.